CLINICAL TRIAL: NCT00940641
Title: A Phase 1, Open, Two Period, Single-Centre, Study to Assess Absorption, Distribution, Metabolism and Excretion (ADME) After Intravenous and 14C-labelled Oral Administration of AZD7325 to Healthy Male Volunteers
Brief Title: Assess the Absorption, Distribution, Metabolism and Excretion of AZD7325 After Intravenous and Oral Administration
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Study withdrawn prior to enrollment due to AZ business decision unrelated to safety.
Sponsor: AstraZeneca (Industry)
Responsible Party: Raj Tummala, M.D./MSD, AstraZeneca
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: D1140C00017
Record Dates: First submitted 2009-07-15; First posted 2009-07-16 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Absorption; Distribution; Metabolism; Excretion
Keywords: Healthy Volunteer
MeSH Terms: interventions — 4-amino-8-(2-fluoro-6-methoxy-phenyl)-N-propylcinnoline-3-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): IV dose of AZD7325
  Interventions: Drug: AZD7325
- 2 (Experimental): 14C oral dose of AZD7325
  Interventions: Drug: AZD7325

INTERVENTIONS:
Drug: AZD7325 — IV Dose
  Arms: 1
Drug: AZD7325 — oral dose
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the absorption, distribution, metabolism and excretion of AZD7325 after intravenous and 14C labeled oral dose

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects Day 1
* Body Mass Index (BMI) > 18 and < 30kg/m2

Exclusion Criteria:

* Clinically relevant disease and abnormalities (past or present) which in the opinion of the investigator, may either put the subject at risk to participate in this study or may influence the results of the study or the subject's ability to participate in the study
* Use of prescription medication within 14 days of the first dose of the investigational product
* Blood loss in excess of 200 mL within 30 days of Day-1 in excess of 500 mL within 90 days of Day-1 or in excess of 1350 mL within 1 year of Day-1 or donation of blood products within 14 days of Day -1

Ages: 35 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2009-08; Primary Completion 2009-10 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
To assess absorption, distribution, metabolism and excretion of AZD7325 after IV dose and 14C oral dose administration | Daily

SECONDARY OUTCOMES:
To evaluate safety and tolerability after a single oral administration of [14C] AZD7325 and after a single intravenous administration of non radio-labelled AZD7325 | Daily

CONTACTS AND LOCATIONS:
Overall Officials: Raj Chetty, MBBS, MD, FRCPath., Principal Investigator — AstraZeneca Alderly Park CPU
Locations (1):
- Research Site, Alderley Park, United Kingdom